CLINICAL TRIAL: NCT00915434
Title: A Single-Dose, Open-Label, Randomized, 4-Way Crossover Study to Characterize the Pharmacokinetics and the Effect of Food of JNJ-31001074 in Healthy Subjects
Brief Title: A Study to Characterize the Pharmacokinetics and Effect of Food on JNJ-31001074 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Clinical Leader, Psychiatry, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CR016180
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: Healthy; Pharmacokinetics
Keywords: Healthy volunteer; Phase I; Non-childbearing potential; JNJ-31001074; Food; Pharmacokinetics
MeSH Terms: interventions — bavisant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: JNJ-31001074

SUMMARY:
This is an open-label (both the physician and healthy volunteer know which treatment will be administered), single-dose, 4-period study to characterize the pharmacokinetics (process by which JNJ-31001074 is absorbed, distributed, metabolized, and eliminated by the body) and effect of food on the pharmacokinetics of JNJ-31001074. The study consists of three phases: a screening phase to determine eligibility, an open-label 4-period treatment phase and an end-of-study/early withdrawal assessment phase.

DETAILED DESCRIPTION:
This is an open-label (both the physician and healthy volunteer know which treatment will be administered), randomized (treatment order determined by chance), single-dose study to characterize the pharmacokinetics (process by which JNJ-31001074 is absorbed, distributed, metabolized, and eliminated by the body) and effect of food on the pharmacokinetics of JNJ-31001074. The study consists of three phases: a screening phase to determine eligibility, an open-label treatment phase and an end-of-study/early withdrawal assessment phase. During the screening phase, healthy volunteers will be evaluated to see if they meet selection criteria as specified in the protocol. Healthy volunteers who meet these criteria will report to the study center on Day -1 to begin treatment. The open-label treatment phase will consist of 4 periods. In each period, volunteers will receive one of the following treatments: Treatment A 1 mg JNJ-31001074, Treatment B 3 mg JNJ-31001074, Treatment C 10 mg JNJ-31001074, and Treatment D 10 mg JNJ-31001074. Treatment A, B and C will be administered under fasting conditions (no food or beverages for 10 hours prior to dosing) and Treatment D will be administered after a high-fat meal. The order in which volunteers will receive each treatment will be determined in a random fashion (like flipping a coin). Each treatment will be separated by a 7-14 day washout period. Multiple blood and urine samples will be collected for 72 hours after each dose. Safety and tolerability will be assessed throughout the volunteer's participation. Volunteers will be instructed to report any adverse events that occur up to 30 days after their last dose of study drug. The maximum study duration for each volunteer is expected to be 66 days. JNJ-31001074 1, 3 or 10 mg will be administered orally on Day 1 of each of the 4 treatment periods (dose depends on participant's treatment sequence)

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer between the ages of 18-55
* if a woman, must be of non childbearing potential (ie, post menopausal or surgically sterile) and have a negative pregnancy test
* body mass index between 18-30
* body weight greater than or equal to 50 kilograms
* blood pressure between 90 and 140 mgHg systolic and no higher than 90 mgHg diastolic
* nonsmoker

Exclusion Criteria:

* History of or current clinically significant medical illness
* clinically significant abnormal laboratory value(s)
* clinically significant abnormal physical examination, vital signs or electrocardiogram
* pregnant, lactating or completed last term pregnancy within six months of screening
* use of any prescription or non prescription medication except for paracetamol (acetaminophen/TYLENOL)
* history of drug or alcohol abuse
* history of smoking or use of nicotine-containing substances within the previous two months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06; Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To characterize the pharmacokinetics of JNJ-31001074 after single-dose administration of 1, 3 and 10 mg JNJ-31001074 and to quantify the effect of food on the pharmacokinetics of 10 mg JNJ-31001074. | Multiple blood and urine samples will be collected for 72 hours after dosing of JNJ-31001074 in each of the 4 treatment periods

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of JNJ-31001074 | up to 66 days (including 21 day screening period)
To assess pharmacokinetic dose proportionality of JNJ-31001074 after single-dose administration of 1, 3 and 10 mg | up to 66 days (including 21 day screening period)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.